CLINICAL TRIAL: NCT04667507
Title: The Pharmacokinetics of Aqueous Dexamethasone and the Inflammatory Cytokine Response After Treatment with a Dexamethasone Intracanalicular Insert - the CYTODEX Study
Brief Title: Pharmacokinetics of Aqueous Dexamethasone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Frank A. Bucci, Jr., M.D. (Other)
Responsible Party: Sponsor-Investigator, Frank A. Bucci, Jr., M.D., Medical Director, Bucci Laser Vision Institute
Organization: Bucci Laser Vision Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-CYTODEX
Record Dates: First submitted 2020-09-21; First posted 2020-12-14 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2022-10

CONDITIONS: Pharmacokinetics; Aqueous Dexamethasone; Inflammatory Cytokine Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Dextenza (Group A) (Experimental): Dextenza (dexamethasone ophthalmic insert 0.4mg) 1-3 days prior to cataract surgery
  Interventions: Drug: Dexamethasone Ophthalmic implant
- Dextenza (Group B) (Experimental): Dextenza (dexamethasone ophthalmic insert 0.4mg) 6-8 days prior to surgery
  Interventions: Drug: Dexamethasone Ophthalmic implant
- Dextenza (Group C) (Experimental): Dextenza (dexamethasone ophthalmic insert 0.4mg) 13-15 days prior to surgery
  Interventions: Drug: Dexamethasone Ophthalmic implant
- Dextenza (Group D) (Experimental): Dextenza (dexamethasone ophthalmic insert 0.4mg) 19-23days prior to surgery
  Interventions: Drug: Dexamethasone Ophthalmic implant
- Dextenza (Group E) (Experimental): Dextenza (dexamethasone ophthalmic insert 0.4mg) 26-31 days prior to surgery
  Interventions: Drug: Dexamethasone Ophthalmic implant
- Control (No Intervention): Will not receive Dextenza (dexamethasone ophthalmic insert 0.4mg)

INTERVENTIONS:
Drug: Dexamethasone Ophthalmic implant — Dexamethasone ophthalmic insert 0.4 mg for intracanalicular use
  Arms: Dextenza (Group A); Dextenza (Group B); Dextenza (Group C); Dextenza (Group D); Dextenza (Group E)

SUMMARY:
The study is being done to measure the absorption of the DEXTENZA implant and inflammation concentration levels in the eye.

ELIGIBILITY:
Inclusion Criteria:

* Male of female, aged 55 or older
* Scheduled to undergo phacoemulsification with the intraocular lens (IOL) implantation for the treatment of cataract
* Willing to comply with study instructions, agree to make study appointments, and complete the course of the study
* Must sign an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate

Exclusion Criteria:

* Known allergy or contraindication to the test article or its components
* Presence of any ocular abnormality or significant illness that, in the investigator's opinion, could affect the subject's health
* History of any illness that could be expected to interfere with the study
* Any condition that, in the opinion of the investigator, would compromise the well-being of the subject or study
* May not be currently using topical or systemic steroids or NSAIDs during the course of the study or within 4 weeks prior to enrolling in the study other than Dextenza and Omidria
* Subject has active corneal, conjunctival, or canalicular infections, including:
* Epithelial herpes simplex keratitis (dendritic keratitis)
* Vaccini
* Varicella
* Mycobacterial infections
* Fungal diseases of the eye
* Dacryocystitis

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics in Aqueous Humor Samples | Measured 1-3 days, 6-8 days, 13-15 days, 19-23 days, and 26-31 days after Dextenza insertion
  Concentration of dexamethasone in the aqueous humor will be determined by an independent laboratory using standardized high-pressure liquid chromatography and mass spectrometry assasys. Pharmacokinetic parameters determined from aqueous humor concentration will minimally include maximum concentration (Cmax).
Pharmacokinetics in Aqueous Humor Samples | Measured 1-3 days, 6-8 days, 13-15 days, 19-23 days, and 26-31 days after Dextenza insertion
  Concentration of inflammatory cytokines (IL-1 beta, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12 (p70), IL-13, TNF alpha, and IFN gamma) in the aqueous humor will be determined by an independent laboratory using standardized high-pressure liquid chromatography and mass spectrometry assasys. Pharmacokinetic parameters determined from aqueous humor concentration will minimally include maximum concentration (Cmax).

SECONDARY OUTCOMES:
Correlation between dexamethasone levels and inflammatory cytokines | 1-3 days, 6-8 days, 13-15 days, 19-23, or 26-31 days after Dextenza insertion
  Test for statistically significant correlations between the aqueous concentrations of dexamethasone and inflammatory cytokines (IL-1 beta, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12 (p70), IL-13, TNF alpha, and IFN gamma) over time

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Bucci, Jr., MD, Principal Investigator — Bucci Laser Vision Institute
Locations (1):
- Bucci Laser Vision, Wilkes-Barre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No